CLINICAL TRIAL: NCT02461602
Title: Eliminate Thromboembolism (ELITE): Improving Anticoagulation in Non-valvular Atrial Fibrillation Patients
Brief Title: Eliminate Thromboembolism: Improving Anticoagulation in Non-valvular Atrial Fibrillation Patients
Acronym: ELITE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00061054
Record Dates: First submitted 2015-05-20; First posted 2015-06-03 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
Keywords: Warfarin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
ELITE (Eliminate Thromboembolism: Improving Anticoagulation in Non-valvular Atrial Fibrillation Patients) is a two year research project to assess warfarin management issues faced by atrial fibrillation (AF) patients in ambulatory settings.

DETAILED DESCRIPTION:
ELITE will be a prospective, multicenter observational study of 500 participants to characterize demographics, comorbidities, risk profiles, socioeconomic status, and patient preferences related to anticoagulation management. The primary study endpoint will be warfarin discontinuation without resumption as documented in the medical record. Secondary outcomes of interest include warfarin adherence and factors associated with suboptimal adherence and/or permanent discontinuation. Clinical data, including demographics, medical history, and comorbidities, will be abstracted and entered by site coordinators. An internal survey developed by Duke Clinical Research Institute (DCRI) will be administered to patients during regularly scheduled clinic visits. Survey items will include patient treatment priorities, perceived risk of bleeding and/or stroke, barriers to adherence, and treatment satisfaction. Subjects will complete a survey at baseline and at the followup visit closest to 6 months after enrollment.

This study will provide the foundation for numerous potential future questions about medication adherence and barriers to treatment, such as a survey on physician preferences/ shared decision-making (concordance between physician and patient preferences), followup to capture clinical events, and interventions to improve long-term medication adherence in AF.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of enrollment
* Electrocardiographically confirmed AF
* Able to complete patient-reported outcomes surveys
* Initiated warfarin therapy in the prior 3 months
* Ability to adhere to regular clinical visits
* Ability to sign informed consent
* Ability to read/comprehend/speak English

Exclusion Criteria:

* Anticipated life expectancy less than six months (as determined by the site investigator)
* Transient AF secondary to a reversible condition (hyperthyroidism, pulmonary embolism, post-cardiothoracic surgery)
* Recent Deep Venous Thrombosis(DVT) or Pulmonary Embolism (PE) (within 6 months)
* Participation in a randomized trial of anticoagulation for AF
* Use of a home international normalized ratio (INR) monitoring system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial Fibrillation patients
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Reason(s) for Warfarin discontinuation | 6 months
Change in Warfarin adherence | Baseline and 6 months

SECONDARY OUTCOMES:
Frequency of hospitalizations | Baseline and 6 months
Frequency of bleeding events | Baseline and 6 months
Change in INR values | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily O'Brien, PhD, Principal Investigator — DCRI
Locations (21):
- United States (21):
  - Foothill Cardiology, Pasadena, California
  - Holy Cross Medical Group, Coral Springs, Florida
  - Charlotte Heart Group, Port Charlotte, Florida
  - Atlanta Institute for Medical Research, Inc., Atlanta, Georgia
  - Atlanta Heart Specialists, Cumming, Georgia
  - Cardiovascular Research of Northwest Indiana, L.L.C., Munster, Indiana
  - Research Integrity, LLC., Owensboro, Kentucky
  - Ochsner Health System, New Orleans, Louisiana
  - Penobscot Bay Medical Center, Rockport, Maine
  - Endeavor Medical Research, Alpena, Michigan
  - Great Lakes Heart and Vascular Institute, Saint Joseph, Michigan
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Duke Cardiology of Lumberton, Lumberton, North Carolina
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Columbia Heart Clinic, PA, Columbia, South Carolina
  - North Texas Research Associates, Allen, Texas
  - Providence Health Center, Waco, Texas
  - Riverside Cardiology Specialists, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No